CLINICAL TRIAL: NCT04601441
Title: Phase 4 Study of Exploring Circulating Tumor DNA (ctDNA) of Metastatic Castration-sensitive Prostate Cancer (mCSPC) Patients Receiving Apalutamide in Japan
Brief Title: Study to Evaluate ctDNA of mCSPC Patients Receiving Apalutamide in Japan
Acronym: CUARTET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kindai University (Other)
Collaborators: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Principal Investigator, Hirotsugu Uemura, Professor, Kindai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 56021927PCR4013; jRCTs071200040 (Registry Identifier: Japan Registry of Clinical Trial (jRCT)); 56021927PCR4013 (Other Grant/Funding Number: Janssen Pharmaceutical K.K.)
Record Dates: First submitted 2020-10-12; First posted 2020-10-23 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Castration-sensitive Prostate Cancer
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apalutamide (Other): Apalutamide 240 mg administered orally once a day as four 60 mg tablets
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Apalutamide 240 mg administered orally once a day as four 60 mg tablets

SUMMARY:
To evaluate changes in genomic alterations for 73 PC driver genes during apalutamide treatment

DETAILED DESCRIPTION:
This clinical study is an open-label, multicenter, interventional, Phase 4 study to evaluate changes in genomic alterations for 73 PC driver genes during apalutamide treatment in patients with mCSPC. A total of 100 participants to be treated by apalutamide will be registered in this study. All participants will undergo blood collection for ctDNA, single-nucleotide polymorphisms (SNPs), and human-leukocyte antigen (HLA) typing at pre- and posttreatment of apalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥20 years.
* Participant has documented diagnosis of metastatic PC with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology.
* Participant has metastatic PC that is castration naïve or castration sensitive and is permitted to receive less than 6-months ADT or CAB before registration and less than 36-months neoadjuvant or adjuvant hormonal therapy.
* If a participant is treated with ADT or CAB, he has maintained a response to hormonal therapy of stable disease or better, by investigator assessment of imaging and PSA.
* Participant is willing to receive apalutamide for mCSPC in the participating site of this study.
* Participant is of Japanese nationality.
* Participant must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

* Participant does not agree to assess ctDNA including 73 PC driver genes, SNPs, and HLA typing.
* Participant has received any prior therapy of abiraterone, docetaxel, enzalutamide, apalutamide or darolutamide.
* Participant has known allergies, hypersensitivity, or intolerance to apalutamide or its excipients (refer to the package insert).
* Participant has contraindications to the use of ADT based on routine treatment.
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the evaluation of active double cancer, etc.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in genomic alterations of 73 PC driver genes between pre- and posttreatment of apalutamide. | Three years or more, 4.5 years or less
  Seventy-three PC driver genes from ctDNA including ARID1A, HSD3B1, MDM4, AKT3, MSH2, MSH6, ERCC3, NFE2L2, IDH1, FANCD2, MLH1, CTNNB1, FOXP1, RYBP, PIK3CB, ATR, PIK3CA, FBXW7, PIK3R1, CHD1, APC, FANCE, CDK6, MET, BRAF, CUL1, KMT2C, NKX3-1, CLU, NCOA2, MYC, CDKN2A, FANCG, FANCC, PTEN, FANCF, CCND1, ATM, ZBTB16, CDKN1B, KRAS, KMT2D, CDK4, MDM2, BRCA2, RB1, ERCC5, FOXA1, RAD51B, AKT1, IDH2, ERCC4, ZFHX3, FANCA, TP53, CDK12, BRCA1, SPOP, RNF43, RAD51C, AKT2, ERCC2, ERCC1, ASXL1, GNAS, RUNX1, ERG, TMPRSS2, KDM6A, AR, MED12, SMARCA1, and PALB2.

SECONDARY OUTCOMES:
The proportion of participants who achieve nadir PSA ≤0.2 ng/mL stratified by baseline genomic alterations for 73 PC driver genes | Three years or more, 4.5 years or less
  The proportion of participants who achieve nadir PSA ≤0.2 ng/mL is defined as the proportion of participants who achieve nadir PSA less than 0.2 ng/mL from apalutamide initiation.
PSA-PFS stratified by baseline genomic alterations for 73 PC driver genes | Three years or more, 4.5 years or less
  The PSA-PFS is defined as the duration from apalutamide initiation to either PSA progression or death, whichever occurs first. The PSA progression will be determined according to the PCWG3 criteria.
PFS stratified by baseline genomic alterations for 73 PC driver genes | Three years or more, 4.5 years or less
  The PFS is defined as the duration from apalutamide initiation to either radiographic progression, clinical progression or death, whichever occurs first. The radiographic and clinical progression will be determined by an investigator's discretion.
OS stratified by baseline genomic alterations for 73 PC driver genes | Three years or more, 4.5 years or less
  The OS is defined as the duration from apalutamide initiation to any death.
Time to CRPC stratified by baseline genomic alterations for 73 PC driver genes | Three years or more, 4.5 years or less
  The time to CRPC is defined as the duration from apalutamide initiation to developing CRPC. The CRPC will be determined according to European Association of Urology (EAU) guidelines 2019.
PFS2 stratified by baseline genomic alterations for 73 PC driver genes | Three years or more, 4.5 years or less
  The PFS2 is defined as the duration from apalutamide initiation to disease progression (PSA progression, radiographic progression, or clinical progression) on the first subsequent therapy for prostate cancer, whichever occurred first. The PSA progression will be determined according to the PCWG3 criteria. The radiographic and clinical progression will be determined by an investigator's discretion.
Safety in the usual clinical practice based on adverse events | From apalutamide initiation to 30 days after the last dose
  Safety observational period is defined as the treatment phase in this study. Adverse events that occur within 30 days after the last dose of apalutamide will be collected, except for lost to follow-up, death, or withdrawal of consent for study participation. For each adverse event, the percentage of participants who experience at least 1 occurrence of the given event will be summarized.
Safety in the usual clinical practice based on potential skin rash events | From apalutamide initiation to 30 days after the last dose
  Safety observational period is defined as the treatment phase in this study. Potential skin rash events that occur within 30 days after the last dose of apalutamide will be collected, except for lost to follow-up, death, or withdrawal of consent for study participation. The percentage of participants who experience at least 1 occurrence of the given event will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Hirotsugu Uemura, MD, PhD, Study Chair — Department of Urology, Kindai University Faculty of Medicine
Locations (1):
- Kindai University Hospital, Ōsaka-sayama, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No